CLINICAL TRIAL: NCT04863716
Title: Effects of Erector Spinae Plane Block on Opioid Consumption in Renal Transplantation Donors
Brief Title: Erector Spinae Plane Block in Renal Transplantation Donors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koc University Hospital (Other)
Responsible Party: Principal Investigator, Özlem Özkalaycı, Anesthesiologist, Koc University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KocUniversityH
Record Dates: First submitted 2021-04-20; First posted 2021-04-28 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Renal Transplantation; Laparoscopic Nephrectomy; Erector Spinae Plane Block
Keywords: Laparoscopic Nephrectomy; Erector Spinae Plane Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane Block (Active Comparator): Erector Spinae Plane Block will be administered to this group.
  Interventions: Procedure: Erector Spinae Plane Block; Procedure: Intravenous fentanyl patient control device
- Control Group (Active Comparator): No regional anesthesia technique will be applied to the control group.
  Interventions: Procedure: Intravenous fentanyl patient control device

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — Erector Spinae Plane Block will be administered before the surgery.
  Arms: Erector Spinae Plane Block
Procedure: Intravenous fentanyl patient control device — 24-hour fentanyl consumption will be recorded.

SUMMARY:
Erector Spina Plan Block (ESPB) is a relatively new, easy-to-apply and safe regional anesthesia technique used to provide postoperative analgesia in various surgeries. Studies showing the clinical benefits of Erector Spina Plan block in renal transplantation surgery are limited to case reports. In this study, the effect of Erector Spina Plan Block on opioid consumption in postoperative period on donor patients who will undergo laparoscopic nephrectomy in renal transplantation surgery will be examined prospectively.

The aim of the study is to provide analgesia to donor patients using less opioids by Erector Spina Plan Block and provide enhanced recovery.

ELIGIBILITY:
Inclusion Criteria:

* Donor patients scheduled for elective nephrectomy in renal transplantation surgery
* ASA I-II
* Patients who are aged between 18-75

Exclusion Criteria:

* Skin infection at the Erector Spina Plan Block area
* Coagulation disorder or using anticoagulant drugs
* End-stage organ and system failure
* Severe pulmonary and/or cardiovascular problems
* Substance addiction or known psychiatric or mental problems
* Chronic painkiller usage

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2022-04-10 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Fentanyl consumption | Postoperative 24 hours
  The amount of fentanyl required by the patient and given by the device will be recorded for the first 24 hours.

SECONDARY OUTCOMES:
Visual Analog Scale | Postoperative 24 hours
  Pain of patients will be evaluated and recorded according to the Visual Analog Scale.
Modified Aldrete Score | Postoperative 1 hour
  Modified Aldrete Score will be used in patient recovery, and scores will be recorded at 5 minute intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- Koç University Hospital, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No